CLINICAL TRIAL: NCT06004843
Title: The Effects of Remimazolam on the Incidence of Hypoxia During Sedated Hysteroscopy for Assisted Reproduction in Overweight or Obese Patients: a Randomized, Controlled Clinical Trial
Brief Title: The Effects of Remimazolam on the Incidence of Hypoxia During Sedated Hysteroscopy for Assisted Reproduction in Overweight or Obese Patients
Acronym: EROP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, diansan su, Vice chair of the department of anesthesiology, RenJi Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: LY2023-115-A
Record Dates: First submitted 2023-08-16; First posted 2023-08-22 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Hypoxia; Hysteroscopy; Overweight or Obesity
Keywords: hypoxia; hysteroscopy; Overweight or Obesity; remimazolam; propofol
MeSH Terms: conditions — Hypoxia; Overweight; Obesity | interventions — remimazolam; Propofol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Remimazolam (Experimental): In this group, participants are sedated with remimazolam and remifentanil.
  Interventions: Drug: remimazolam
- propofol (Active Comparator): In this group, participants are sedated with propofol and remifentanil.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: remimazolam — in this group,patients are treated with remimazolam and remifentanil for reduced sedation.
  Arms: Remimazolam
Drug: Propofol — in this group,patients are treated with propofol and remifentanil for reduced sedation.
  Arms: propofol

SUMMARY:
Hypoxia is a common adverse event during sedated hysteroscopy for assisted reproduction, and it is more likely to occur in overweight or obese patients. In sedated gastroscopy, the incidence of hypoxia with remimazolam is lower than that with propofol. The present study is a single-center, randomized, single-blind, controlled clinical trial. Overweight or obese patients undergoing sedated hysteroscopy for diagnosis and treatment, with ASA grade I or II, were selected as subjects and randomly divided into an experimental group and a control group, with 300 subjects in each group. Sedation induction and maintenance are performed using remimazolam or propofol combined with remifentanil, respectively, to compare the incidence of hypoxia during surgery between the two groups of patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 20 and 50 years.
2. Patients undergoing sedated hysteroscopy for assisted reproduction.
3. ASA classification I-II.
4. BMI ≥ 23 kg/㎡.
5. Patients who have signed an informed consent form.

Exclusion Criteria:

1. SpO2 < 95% in patients inhaling air upon entering the room.
2. Diagnosed with chronic obstructive pulmonary disease (COPD) or currently suffering from other acute and chronic lung diseases requiring long-term or intermittent oxygen therapy.
3. Patients with a history of mental and neurological disorders: such as depression, severe central nervous system depression, Parkinson's disease, basal ganglia disease, schizophrenia, epilepsy, Alzheimer's disease, myasthenia gravis, etc.
4. Patients with severe liver dysfunction.
5. Patients with severe renal insufficiency (requiring dialysis before surgery).
6. Severe heart failure (METS < 4).
7. History of drug abuse and/or alcohol abuse within the 2 years preceding the screening period (consuming more than three times the standard alcoholic beverages daily, approximately 10g of alcohol, or equivalent to 50g of Chinese alcohol).
8. Allergies or contraindications to benzodiazepines, flumazenil, opiates and their rescue medications, propofol, eggs, or soy products.
9. Breastfeeding women.
10. Patients whom investigator believe are unsuitable for participating in this trial.

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 600 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
The incidence of hypoxia | Participants will be followed for the duration of their hospital stay, with an expected average of about 2 hours.
  75%≤ SpO2% ≤89% for<60s

SECONDARY OUTCOMES:
The incidence of sub-clinical respiratory depression | Participants will be followed for the duration of their hospital stay, with an expected average of about 2 hours.
  90%≤ SpO2<95%
The incidence of severe hypoxia | Participants will be followed for the duration of their hospital stay, with an expected average of about 2 hours.
  SpO2<75% or 75%≤ SpO2≤89% for≥60s
The incidence of other adverse events | Participants will be followed for the duration of their hospital stay, with an expected average of about 2 hours.
  Other adverse events recorded by tools proposed by the World Society of Intravenous Anesthesia International Sedation Task Force

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital, Shanghai, Pudong New Area, China

IPD SHARING:
Plan to Share IPD: No